CLINICAL TRIAL: NCT06333951
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 193 Alone or in Combination With Other Therapies in Subjects With Advanced Thoracic Tumors With Homozygous MTAP-deletion (Master Protocol)
Brief Title: AMG 193 Alone or in Combination With Other Therapies in Subjects With Advanced Thoracic Tumors With Homozygous MTAP-deletion (Master Protocol) (MTAPESTRY 104).
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230167
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Tumors; Non-small Cell Lung Cancer
Keywords: Oncology; Methylthioadenosine phosphorylase; AMG 193; PRMT5 inhibitor; MTAP; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Carboplatin; Paclitaxel; pembrolizumab; Pemetrexed; sotorasib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Subprotocol A: Non-Small Cell Lung Cancer (NSCLC) Arm A (Experimental): Participants with MTAP-deleted NSCLC will receive a regimen of AMG 193 orally (PO) and carboplatin, paclitaxel, and pembrolizumab intravenously (IV)
  Interventions: Drug: AMG 193; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pembrolizumab
- Subprotocol A: NSCLC Arm B (Experimental): Participants with MTAP-deleted NSCLC will receive a regimen of AMG 193 PO and carboplatin, pemetrexed, and pembrolizumab IV
  Interventions: Drug: AMG 193; Drug: Carboplatin; Drug: Pembrolizumab; Drug: Pemetrexed
- Subprotocol A: NSCLC Arm C (Experimental): Participants with MTAP-deleted NSCLC will receive a combination of AMG 193 PO and pembrolizumab IV
  Interventions: Drug: AMG 193; Drug: Pembrolizumab
- Subprotocol B: NSCLC With KRasG12C Mutation (Experimental): Participants with MTAP-deleted NSCLC and KRasG12C mutation will receive a combination of AMG 193 and sotorasib PO
  Interventions: Drug: AMG 193; Drug: Sotorasib
- Subprotocol C: NSCLC With Brain Metastases (Experimental): Participants with MTAP-deleted NSCLC with brain metastases will receive AMG 193 PO
  Interventions: Drug: AMG 193

INTERVENTIONS:
Drug: AMG 193 — Administered PO
Drug: Carboplatin — Administered IV
  Arms: Subprotocol A: NSCLC Arm B; Subprotocol A: Non-Small Cell Lung Cancer (NSCLC) Arm A
Drug: Paclitaxel — Administered IV
  Arms: Subprotocol A: Non-Small Cell Lung Cancer (NSCLC) Arm A
Drug: Pembrolizumab — Administered IV
  Arms: Subprotocol A: NSCLC Arm B; Subprotocol A: NSCLC Arm C; Subprotocol A: Non-Small Cell Lung Cancer (NSCLC) Arm A
Drug: Pemetrexed — Administered IV
  Arms: Subprotocol A: NSCLC Arm B
Drug: Sotorasib — Administered PO
  Arms: Subprotocol B: NSCLC With KRasG12C Mutation

SUMMARY:
The study aims to determine maximum tolerated dose (MTD) or recommended combination dose of the MTA-cooperative PRMT5 inhibitor AMG 193 administered in combination with other therapies in adult participants with metastatic or locally advanced methylthioadenosine phosphorylase (MTAP)-deleted thoracic tumors. The study also aims to determine the safety profile of AMG 193 administered in combination with other therapies in adult participants with metastatic or locally advanced MTAP-deleted thoracic tumors.

ELIGIBILITY:
Inclusion Criteria

Subprotocol A, B, and C

* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years).
* Tumor tissue (formalin-fixed, paraffin-embedded sample) or an archival block must be available. Participants without archived tumor tissue available may be allowed to enroll by undergoing tumor biopsy before AMG 193 dosing.
* Homozygous MTAP-deletion
* Able to swallow and retain PO administered study treatment.
* Disease measurable as defined by RECIST v1.1.

Subprotocol A - Histologically or cytologically confirmed diagnosis of NSCLC.

Arm A (AMG 193 + carboplatin + paclitaxel + pembrolizumab):

- Predominantly squamous histology.

Arm B (AMG 193 + carboplatin + pemetrexed + pembrolizumab):

- Predominantly non-squamous histology.

Arm C (AMG 193 + pembrolizumab):

- PD-L1 positive.

Subprotocol B - Histologically confirmed NSCLC with homozygous MTAP-deletion and KRAS p.G12C mutation.

Subprotocol C

* Histologically or cytologically confirmed diagnosis of NSCLC with brain metastases.
* Brain lesion meeting RANO-BM criteria for measurable disease.

Exclusion Criteria

Subprotocol A, B, and C

* Cardiovascular and pulmonary exclusion criteria as defined in the protocol.
* Gastrointestinal tract disease causing the inability to take PO medication, malabsorption syndrome, requirement for IV alimentation, gastric/jejunal tube feeds, uncontrolled inflammatory gastrointestinal disease (eg, Crohn's disease, ulcerative colitis).
* History of solid organ transplant.
* Major surgery within 28 days of first dose of AMG 193.
* Prior treatment with a MAT2A inhibitor or a PRMT5 inhibitor.
* Radiation therapy within 28 days of first dose.

Subprotocol A

- Autoimmune disease or immunodeficiency disease as defined in the protocol'

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2028-10-27 (Estimated); Study Completion 2031-10-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose Limiting Toxicities (DLT) | Up to approximately 21 days
Number of Participants Experiencing Treatment Emergent Adverse Events (TEAE) | Up to approximately 3 years
  TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs. A serious TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s) that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Number of Participants Experiencing Serious Adverse Events (SAE) | Up to approximately 3 years
  An SAE is defined as any AE that results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect or important medical events that do not meet the preceding criteria but based on appropriate medical judgment may jeopardize the participant or may require medical or surgical intervention to prevent any of the outcomes listed above.

SECONDARY OUTCOMES:
Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to approximately 3 years
Disease Control (DC) per RECIST v1.1 | Up to approximately 3 years
Duration of Response (DOR) per RECIST v1.1 | Up to approximately 3 years
Time to Response (TTR) per RECIST v1.1 | Up to approximately 3 years
Overall Survival (OS) per RECIST v1.1 | Up to approximately 3 years
Progression-free Survival (PFS) per RECIST v1.1 | Up to approximately 3 years
Maximum Plasma Concentration (Cmax) of AMG 193 | Up to Day 1 of Cycle 5 (one cycle = 21 days)
Time to Maximum Plasma Concentration (tmax) of AMG 193 | Up to Day 1 of Cycle 5 (one cycle = 21 days)
Area Under the Plasma Concentration-time Curve (AUC) of AMG 193 | Up to Day 1 of Cycle 5 (one cycle = 21 days)
Intracranial objective response (IOR) per Response Assessment in Neuro Oncology Brain Metastases (RANO-BM ) | Up to approximately 3 years
Intracranial Disease Control (IDC) per RANO-BM | Up to approximately 3 years
Intracranial Duration of Response (IDOR) per RANO-BM | Up to approximately 3 years
Time to Intracranial Radiation Therapy per RANO-BM | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (83):
- United States (26):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Duarte, California
  - Translational Research in Oncology US Inc, Trio Central Pharmacy, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of California Los Angeles, Santa Monica, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - HealthPartners Institute, Saint Paul, Minnesota
  - Saint Lukes Hospital of Kansas City, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Grossman School of Medicine, New York, New York
  - Perlmutter Cancer Center at New York University Langone Hospital----Long Island, New York, New York
  - Upstate University Hospital, Syracuse, New York
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - Texas Oncology - Dallas Fort Worth, Dallas, Texas
  - US Oncology Research Investigational Products Center, Dallas, Texas
  - Oncology Consultants Cancer Center, Houston, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists PC, Fairfax, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Argentina (3):
  - Instituto Argentino de Diagnóstico y Tratamiento, Ciudad Automona de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Cemic, Ciudad Autonoma Buenos Aires
- Australia (2):
  - Orange Health Service, Orange, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
- Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège, Belgium
- Brazil (5):
  - Oncosite Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Cipo - Centro Integrado de Pesquisa em Oncologia, Porto Alegre, Rio Grande do Sul
  - Fund Faculdade Regional Med Sao Jose Rio Preto, São José do Rio Preto, São Paulo
  - Beneficencia Portuguesa de Sao Paulo - Bp, São Paulo, São Paulo
  - Instituto Cancer Sao Paulo Icesp, São Paulo
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- China (7):
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jilin Cancer Hospital, Changchun, Jilin
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Beijing Cancer Hospital, Beijing
- France (4):
  - Institut Bergonie, Bordeaux
  - Hopital de la Timone, Marseille
  - Institut de Cancerologie de l Ouest Rene Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - Alexandra Hospital, Athens
  - Saint Luke Hospital, Thessaloniki
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Alessandria
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano (MI)
  - Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona
- Japan (4):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Gliwice
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (3):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of reevaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com